CLINICAL TRIAL: NCT03097484
Title: The Effect of Aromatherapy on Neonatal Abstinence Syndrome and Salivary Cortisol Levels
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: John M. Daniel (Other)
Responsible Party: Sponsor-Investigator, John M. Daniel, Fellow, Department of Pediatrics, Division of Neonatology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0159-F2L
Record Dates: First submitted 2017-03-15; First posted 2017-03-31 (Actual); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Neonatal Abstinence Syndrome; Aromatherapy
MeSH Terms: conditions — Neonatal Abstinence Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard therapy plus Aromatherapy (Experimental): These infants will receive aromatherapy, consisting of Lavender and Chamomile essential oils, in addition to standard care, which includes morphine replacement therapy, infant massage, PT, OT, and music therapy.
  Interventions: Drug: lavender and chamomile essential oils
- Standard therapy ALONE (No Intervention): These infants receive standard care ONLY, which includes morphine replacement therapy, infant massage, PT, OT, and music therapy.

INTERVENTIONS:
Drug: lavender and chamomile essential oils — Our patches are obtained from BioEsse Technologies™. Each patch contains a 50:50 mixture of Lavender and Chamomile essential oils in a 55 microliter standard dose patch. The patches release the aromatherapy over a 2-8 hours period and the diffusion rate of each patch is identical. The back of the patch is layered with a hypoallergenic medical grade adhesive, similar to the material found on ECG leads.
  Other Names: Lavendula, chamomilla
  Arms: Standard therapy plus Aromatherapy

SUMMARY:
Determine the effectiveness of lavender and chamomile aromatherapy of mitigation of symptoms of Neonatal Abstinence Syndrome

DETAILED DESCRIPTION:
The United States, Appalachia, Eastern Kentucky in particular, is in the midst of a major opioid abuse epidemic. This current epidemic is driven by misuse of prescription painkillers, i.e. Subutex and Saboxone. As prescription pills become more expensive and harder to acquire, addicts are seeking similar, cheaper drugs; such as heroin. From 1998 to 2011, the prevalence of opioid abuse and dependence amongst pregnant women has increased by 127%, from 1.7 per 1000 to 3.9 per 1000. Neonatal Abstinence Syndrome (NAS) or neonatal opioid withdrawal syndrome is a condition produces gastrointestinal and autonomic neurologic dysfunction. Infants with severe withdrawal experience dysregulation of autonomic functions, resulting in feeding difficulty, diarrhea, excessive sleepiness, and tremors.Nearly two thirds of all babies exposed to opioids during gestation will require admission to a neonatal intensive care unit for management of withdrawal symptoms. During a typical year the Neonatal Intensive Care Unit (NICU) at Kentucky Children's Hospital admits approximately 100-120 infants exhibiting NAS symptoms; these infants have a typical length of stay of 24 days if they require pharmacologic treatment.

The mainstay of treatment for NAS involves opioid replacement therapy with morphine to minimize withdrawal symptoms. Once symptoms are well controlled, the infant is said to have been "captured." At this point a slow weaning of his morphine dose occurs. The infants' clinical status is assessed with the Finnegan Scoring system, which examines symptoms such as crying, excessive sleepiness or difficulty sleeping, insomnia, or tremors along with objective findings such as temperature and respiratory rate.

In addition to pharmacotherapy, alternative and complementary medicine techniques are slowly entering the NAS treatment algorithm. Treatments such as music therapy infant massage, kangaroo care, aromatherapy, and acupressure are now employed in NICUs in addition to traditional opioids replacement. However, few studies exist in the literature to evaluate their effectiveness.

Aromatherapy is the practice of using natural essential oils to achieve a desired effect in an individual. Scents such as lavender and chamomile have been documented to have a soothing calming effect. Studies involving infants shown that lavender not only reduce crying and enhance sleep, but also reduce levels of salivary cortisol, a stress hormone. Additionally, aromatherapy is currently used as an adjunctive therapy at the University of Kentucky's Markey Cancer Center.

Salivary cortisol is a non-invasive biomarker that has proven useful for monitoring stress in neonates. It is a simple and painless method for monitoring the stress hormone cortisol. Salivary cortisol has been used successfully in infants as a method to assess infant stress associated with prone position versus supine positioning.These studies have shown that salivary cortisol levels vary with stressful or soothing stimuli.

To date, no dangerous or deleterious effects have been described from traditional inhalational use of aromatherapy or with salivary cortisol sampling. Studies have shown aromatherapy to be an effective adjunctive therapy by proving a calming effect. In our patient population it may prove to be a useful complimentary therapy ultimately reducing infant stress, hospital length of stay, and burden of opioid use. Additionally, salivary cortisol's ease of collection and non-invasive nature make it an ideal biomarker to study.

ELIGIBILITY:
Inclusion Criteria:

* Infants greater than or equal to 36 weeks EGA
* Intrauterine opioid exposure
* Primary diagnosis of NAS
* Parental permission to participate

Exclusion Criteria:

* Infants less than 36 weeks EGA
* Major congenital anomalies
* Latrogenic drug withdrawal
* Diagnosis of infection or respiratory distress
* Prior initiation of opioid replacement therapy
* Non-English speaking
* Infants with respiratory conditions

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2015-07-25 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Daniel, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ang JY, Lua JL, Mathur A, Thomas R, Asmar BI, Savasan S, Buck S, Long M, Shankaran S. A randomized placebo-controlled trial of massage therapy on the immune system of preterm infants. Pediatrics. 2012 Dec;130(6):e1549-58. doi: 10.1542/peds.2012-0196. Epub 2012 Nov 12. PMID 23147978
- [Result] Candia MF, Osaku EF, Leite MA, Toccolini B, Costa NL, Teixeira SN, Costa CR, Piana PA, Cristovam MA, Osaku NO. Influence of prone positioning on premature newborn infant stress assessed by means of salivary cortisol measurement: pilot study. Rev Bras Ter Intensiva. 2014 Apr-Jun;26(2):169-75. doi: 10.5935/0103-507x.20140025. PMID 25028952
- [Result] Conde-Agudelo A, Diaz-Rossello JL. Kangaroo mother care to reduce morbidity and mortality in low birthweight infants. Cochrane Database Syst Rev. 2014 Apr 22;(4):CD002771. doi: 10.1002/14651858.CD002771.pub3. PMID 24752403
- [Result] Field T, Diego M, Hernandez-Reif M, Cisneros W, Feijo L, Vera Y, Gil K, Grina D, Claire He Q. Lavender fragrance cleansing gel effects on relaxation. Int J Neurosci. 2005 Feb;115(2):207-22. doi: 10.1080/00207450590519175. PMID 15764002
- [Result] Field T, Field T, Cullen C, Largie S, Diego M, Schanberg S, Kuhn C. Lavender bath oil reduces stress and crying and enhances sleep in very young infants. Early Hum Dev. 2008 Jun;84(6):399-401. doi: 10.1016/j.earlhumdev.2007.10.008. Epub 2007 Nov 28. PMID 18053656
- [Result] Filippelli AC, White LF, Spellman LW, Broderick M, Highfield ES, Sommers E, Gardiner P. Non-Insertive Acupuncture and Neonatal Abstinence Syndrome: A Case Series from an Inner City Safety Net Hospital. Glob Adv Health Med. 2012 Sep;1(4):48-52. doi: 10.7453/gahmj.2012.1.4.007. PMID 24078899
- [Result] Hayes MJ, Brown MS. Epidemic of prescription opiate abuse and neonatal abstinence. JAMA. 2012 May 9;307(18):1974-5. doi: 10.1001/jama.2012.4526. Epub 2012 Apr 30. No abstract available. PMID 22546607
- [Result] Loewy J, Stewart K, Dassler AM, Telsey A, Homel P. The effects of music therapy on vital signs, feeding, and sleep in premature infants. Pediatrics. 2013 May;131(5):902-18. doi: 10.1542/peds.2012-1367. Epub 2013 Apr 15. PMID 23589814
- [Result] Maeda A, Bateman BT, Clancy CR, Creanga AA, Leffert LR. Opioid abuse and dependence during pregnancy: temporal trends and obstetrical outcomes. Anesthesiology. 2014 Dec;121(6):1158-65. doi: 10.1097/ALN.0000000000000472. PMID 25405293
- [Result] Namazi M, Amir Ali Akbari S, Mojab F, Talebi A, Alavi Majd H, Jannesari S. Aromatherapy with citrus aurantium oil and anxiety during the first stage of labor. Iran Red Crescent Med J. 2014 Jun;16(6):e18371. doi: 10.5812/ircmj.18371. Epub 2014 Jun 5. PMID 25068058
- [Result] Olson SL. Bedside musical care: applications in pregnancy, childbirth, and neonatal care. J Obstet Gynecol Neonatal Nurs. 1998 Sep-Oct;27(5):569-75. doi: 10.1111/j.1552-6909.1998.tb02624.x. PMID 9773369
- [Result] Parlier AB, Fagan B, Ramage M, Galvin S. Prenatal care, pregnancy outcomes, and postpartum birth control plans among pregnant women with opiate addictions. South Med J. 2014 Nov;107(11):676-83. doi: 10.14423/SMJ.0000000000000189. PMID 25365432
- [Result] Patrick SW, Schumacher RE, Benneyworth BD, Krans EE, McAllister JM, Davis MM. Neonatal abstinence syndrome and associated health care expenditures: United States, 2000-2009. JAMA. 2012 May 9;307(18):1934-40. doi: 10.1001/jama.2012.3951. Epub 2012 Apr 30. PMID 22546608
- [Result] Tang SK, Tse MY. Aromatherapy: does it help to relieve pain, depression, anxiety, and stress in community-dwelling older persons? Biomed Res Int. 2014;2014:430195. doi: 10.1155/2014/430195. Epub 2014 Jul 13. PMID 25114901
- [Result] Thomas DV. Aromatherapy: mythical, magical, or medicinal? Holist Nurs Pract. 2002 Oct;16(5):8-16. doi: 10.1097/00004650-200210000-00005. PMID 12465213
- [Result] Tryphonopoulos PD, Letourneau N, Azar R. Approaches to salivary cortisol collection and analysis in infants. Biol Res Nurs. 2014 Oct;16(4):398-408. doi: 10.1177/1099800413507128. Epub 2013 Oct 16. PMID 24136995
- [Derived] Pahl A, Young L, Buus-Frank ME, Marcellus L, Soll R. Non-pharmacological care for opioid withdrawal in newborns. Cochrane Database Syst Rev. 2020 Dec 21;12(12):CD013217. doi: 10.1002/14651858.CD013217.pub2. PMID 33348423

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Therapy ALONE | Standard Therapy Plus Aromatherapy
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy ALONE | Standard Therapy Plus Aromatherapy | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: days] | 38.14 (9) | 38.86 (5) | 38.50 (7.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 9 | 8 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
Birth Weight [Mean (Standard Deviation); unit: kilograms] | 2.9 (0.5) | 3.1 (0.4) | 3.0 (.45)
Opioid Exposure Only [Count of Participants; unit: Participants] | 8 | 9 | 17
Multi-Drug Exposure [Count of Participants; unit: Participants] | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospitalization
Description: How long the infant remains hospitalized.
Time Frame: Up to 4 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Therapy ALONE | Standard Therapy Plus Aromatherapy
Number analyzed (Participants) | 19 | 19
days | 17.8 (10.1) | 11.4 (6.6)
Statistical Analysis 1: Comparison: Standard Therapy ALONE vs Standard Therapy Plus Aromatherapy; Test type: Superiority; p = 0.03, t-test, 2 sided

2. Secondary Outcome: Length of Medication Therapy
Description: How long the infant requires medication to treat symptoms.
Time Frame: Up to 4 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Therapy ALONE | Standard Therapy Plus Aromatherapy
Number analyzed (Participants) | 19 | 19
days | 12.7 (10.1) | 7.4 (6.1)
Statistical Analysis 1: Comparison: Standard Therapy ALONE vs Standard Therapy Plus Aromatherapy; Test type: Superiority; p = 0.05, t-test, 2 sided — 0.05 is the calculated p-value (not the threshold for statistical significance)

ADVERSE EVENTS:
Time Frame: Until release from the hospital (up to 50 days post-birth)
Description: Data were collected from hospital electronic medical records.
Arm/Group | Standard Therapy ALONE | Standard Therapy Plus Aromatherapy
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

LIMITATIONS AND CAVEATS:
Interpretation is limited by being a single-center, open-label trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT03097484/Prot_SAP_000.pdf